CLINICAL TRIAL: NCT02271932
Title: Multi-institutional Trial of Non-operative Management of Uncomplicated Pediatric Appendicitis
Brief Title: Multi-institutional Trial of Non-operative Management of Appendicitis
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Nationwide Children's Hospital (Other)
Collaborators: Children's Hospital and Health System Foundation, Wisconsin (Other); Comer Children' Hospital (Unknown); C.S. Mott Children's Hospital (Other); James Whitcomb Riley Hospital for Children (Other); Kosair Children' Hospital (Unknown); Ann & Robert H Lurie Children's Hospital of Chicago (Other); St. Louis Children's Hospital (Other); American Family Children's Hospital (Other); Children's Hospital Medical Center, Cincinnati (Other)
Responsible Party: Principal Investigator, Peter Minneci, Assistant Professor of Surgery and Pediatrics, Nationwide Children's Hospital
Other Study IDs: IRB14-00651; 1507-31325 (Other Grant/Funding Number: PCORI)
Record Dates: First submitted 2014-10-20; First posted 2014-10-22 (Estimated); Last update posted 2023-02-09 (Actual); Status verified 2023-02

CONDITIONS: Appendicitis
Keywords: appendicitis; non-operative management; children; pediatric
MeSH Terms: conditions — Appendicitis | interventions — Anti-Bacterial Agents

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Surgery: Surgical management with appendectomy consists of hospital admission with initiation of intravenous antibiotics and urgent appendectomy .
- Non-operative: Non-operative management consists of hospital admission for observation with a minimum of 24 hours of intravenous antibiotics and a minimum of 12 hours nil per os (NPO). With clinical improvement, patients are switched to oral antibiotics and discharged home with a prescription for oral antibiotics to complete a total antibiotic course of 7 days (including the duration of intravenous antibiotics).
  Interventions: Other: Non-operative

INTERVENTIONS:
Other: Non-operative — Patients will receive only antibiotics and will not undergo appendectomy unless they do not improve or their appendicitis recurs
  Other Names: Non-operative management with antibiotics alone
  Groups: Non-operative

SUMMARY:
A successful non-operative management strategy for early appendicitis will decrease the number of children requiring surgery and may improve the quality of care related to the treatment of appendicitis. To account for the child-family perspective and treatment preferences, the investigators will perform a study in which patients and their families choose between antibiotics alone (Non-operative group) or appendectomy (Surgery group) at ten U.S. hospitals. This study will determine the effectiveness of non-operative management of early appendicitis with antibiotics alone in children and compare differences in morbidity, disability, quality of life, satisfaction, and cost between families choosing surgery or non-operative management.

DETAILED DESCRIPTION:
Several randomized controlled trials comparing appendectomy to antibiotics alone in adults with acute appendicitis have been reported from non-U.S. countries. These studies reveal that non-operative management of appendicitis is a safe treatment for appendicitis and is associated with a significantly lower risk of complications than appendectomy. We have recently completed the first study in the U.S. examining the feasibility of non-operative management of uncomplicated appendicitis in children. In our pilot study, patients and their families chose between urgent appendectomy or antibiotics alone for treatment of uncomplicated appendicitis. The success rate of non-operative management was 90% at 30 days and 80% at a median follow-up of 8 months. In addition, patients in the non-operative group demonstrated a significantly faster return to normal activity and reported higher quality of life scores. The current proposal seeks to further investigate the effectiveness of non-operative management with antibiotics alone as a treatment option for children with uncomplicated appendicitis. When randomized trials are not feasible due to strong treatment preferences or when only a small proportion of patients will accept randomization, a parallel group non-randomized study where participants are allocated to their preferred treatment is a valuable alternative. Based on feedback from a multi-disciplinary stakeholder group that was convened to assess the potential impact of family preferences on study outcomes, recruitment, and generalizability, we propose a multi-institutional trial in which patients and their families choose between antibiotics alone (Non-operative group) or appendectomy (Surgery group). We hypothesize that non-operative management will be successful in 75% of patients at 1 year follow-up and will be associated with fewer disability days, higher quality of life scores, and lower costs than appendectomy. This study will enroll 795 patients, age 8-17 years, with uncomplicated appendicitis at 10 children's hospitals. The primary outcomes are: 1) differences in treatment-related disability between non-operative management and surgery in children with uncomplicated appendicitis across 10 children's hospitals; and 2) the success rate of non-operative management of uncomplicated appendicitis at 10 children's hospitals, defined as the percent of patients treated non-operatively who do not undergo an appendectomy. Secondary outcomes include differences between the groups in rates of complicated appendicitis, post-treatment related complications, disability days of the parent, quality of life and healthcare satisfaction measures, and total costs and the incremental cost-effectiveness of non-operative management relative to appendectomy. The proposed study will expand upon our previous pilot study by including patients from both freestanding and non-freestanding children's hospitals with both urban and rural demographies to determine the success rate and morbidity associated with non-operative management in a population that better represents the overall population of children in the U.S. Successful completion of this study may provide evidence for the effectiveness of non-operative management of uncomplicated appendicitis as an alternative first line therapy in children.

ELIGIBILITY:
Inclusion Criteria:

* English and non-English speaking patients
* Age : 8-17 years
* US or CT confirmed early appendicitis with US showing hyperemia, ≤ 1.1 cm in diameter, compressible or non-compressible, no abscess, no fecalith, no phlegmon or CT showing hyperemia, fat stranding, ≤ 1.1 cm in diameter, no abscess, no fecalith, no phlegmon
* White Blood Cell count > 5,000/µL and ≤ 18,000/µL
* Abdominal pain ≤ 48hours prior to receiving antibiotics

Exclusion Criteria:

* History of chronic intermittent abdominal pain
* Pain > 48 hours prior to first antibiotic dose
* Diffuse peritonitis
* Positive urine pregnancy test
* White Blood Cell ≤ 5,000/µL or ≥ 18,000/µL
* Presence of a fecalith on imaging
* Evidence on imaging studies concerning for evolving perforated appendicitis including abscess or phlegmon
* Communication difficulties (e.g. severe developmental delay)

Ages: 8 Years to 17 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Study Population: Children with uncomplicated appendicitis
Sampling Method: Probability Sample
Enrollment: 1076 (Actual)
Dates: Start 2014-10-01 (Actual); Primary Completion 2019-11-01 (Actual); Study Completion 2023-11-01 (Estimated)

PRIMARY OUTCOMES:
Success rate | 1 year
  success rate at 1 year is percent of patients choosing non-operative management who have not undergone an appendectomy
Disability Days | 1 year
  Number of days without normal schedule

SECONDARY OUTCOMES:
Perforated appendicitis | 1 year
  percent of patients with perforated appendicitis at operation

CONTACTS AND LOCATIONS:
Locations (1):
- Nationwide Children's Hospital, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Minneci PC, Sulkowski JP, Nacion KM, Mahida JB, Cooper JN, Moss RL, Deans KJ. Feasibility of a nonoperative management strategy for uncomplicated acute appendicitis in children. J Am Coll Surg. 2014 Aug;219(2):272-9. doi: 10.1016/j.jamcollsurg.2014.02.031. Epub 2014 Apr 13. PMID 24951281
- [Background] Minneci PC, Mahida JB, Lodwick DL, Sulkowski JP, Nacion KM, Cooper JN, Ambeba EJ, Moss RL, Deans KJ. Effectiveness of Patient Choice in Nonoperative vs Surgical Management of Pediatric Uncomplicated Acute Appendicitis. JAMA Surg. 2016 May 1;151(5):408-15. doi: 10.1001/jamasurg.2015.4534. PMID 26676711
- [Background] Gonzalez DO, Deans KJ, Minneci PC. Role of non-operative management in pediatric appendicitis. Semin Pediatr Surg. 2016 Aug;25(4):204-7. doi: 10.1053/j.sempedsurg.2016.05.002. Epub 2016 May 10. PMID 27521709
- [Derived] Gil LA, Asti L, Chen HF, Saito JM, Pattisapu P, Deans KJ, Minneci PC; Midwest Pediatric Surgery Consortium. Cost-Effectiveness of Nonoperative Management vs Upfront Laparoscopic Appendectomy for Pediatric Uncomplicated Appendicitis for 1 Year. J Am Coll Surg. 2025 Mar 1;240(3):288-298. doi: 10.1097/XCS.0000000000001232. Epub 2025 Feb 14. PMID 39560281
- [Derived] Minneci PC, Hade EM, Gil LA, Metzger GA, Saito JM, Mak GZ, Hirschl RB, Gadepalli S, Helmrath MA, Leys CM, Sato TT, Lal DR, Landman MP, Kabre R, Fallat ME, Cooper JN, Deans KJ; Midwest Pediatric Surgery Consortium. Demographic and Clinical Characteristics Associated With the Failure of Nonoperative Management of Uncomplicated Appendicitis in Children: Secondary Analysis of a Nonrandomized Clinical Trial. JAMA Netw Open. 2022 May 2;5(5):e229712. doi: 10.1001/jamanetworkopen.2022.9712. PMID 35499827
- [Derived] Minneci PC, Hade EM, Lawrence AE, Sebastiao YV, Saito JM, Mak GZ, Fox C, Hirschl RB, Gadepalli S, Helmrath MA, Kohler JE, Leys CM, Sato TT, Lal DR, Landman MP, Kabre R, Fallat ME, Cooper JN, Deans KJ; Midwest Pediatric Surgery Consortium. Association of Nonoperative Management Using Antibiotic Therapy vs Laparoscopic Appendectomy With Treatment Success and Disability Days in Children With Uncomplicated Appendicitis. JAMA. 2020 Aug 11;324(6):581-593. doi: 10.1001/jama.2020.10888. PMID 32730561